CLINICAL TRIAL: NCT05487976
Title: A Phase III Clinical Study of the Efficacy and Safety of Recombinant Human Activated Coagulation Factor VII for Injection in Patients With Hemophilia With Inhibitors
Brief Title: Clinical Study of Recombinant Human Activated Coagulation Factor VII for Injection in Patients With Hemophilia With Inhibitor
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQG203-III-01
Record Dates: First submitted 2022-04-11; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Hemophilia A; Hemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recombinant human activated coagulation factor VII for injection (Experimental): Each subject in this study received on-demand treatment with recombinant human activated coagulation factor VII for injection for 24 weeks. The single dose for each bleeding event was 90 μg/kg, and the number of doses was increased according to the remission after treatment.
  Interventions: Drug: Recombinant human activated coagulation factor VII for injection

INTERVENTIONS:
Drug: Recombinant human activated coagulation factor VII for injection — Human coagulation factor VII is a vitamin K-dependent serine endogenous protease, and its activated form plays an important role in the coagulation process. Recombinant human activated coagulation factor VII is an activated state coagulation factor VII obtained by recombinant means.

SUMMARY:
Human coagulation factor VII is a vitamin K-dependent serine endogenous protease, and its activated form plays an important role in the coagulation process. Recombinant human activated coagulation factor VII is an activated state coagulation factor VII obtained by recombinant means.

ELIGIBILITY:
Inclusion Criteria:

* 1 Diagnosed as congenital hemophilia A or B, and meet the following conditions:

  1. FⅧ<1% or FIX activity<2%;
  2. FⅧ inhibitor or FⅨ inhibitor titer in the screening period>5 BU (Nijmegen modified Bethesda method of detection)."
* 2 Age ≥18 and ≤65 years, male or female.
* 3 There have been at least two incidents of bleeding of any kind in the last six months.
* 4 No other drugs for the treatment of hemophilia have been used within 72hours (3 days) before administration, including prothrombin complex and any coagulation factor VII or activated coagulation factor VII、coagulation factor VIII、coagulation factor IX products, cryoprecipitate, fresh plasma and whole blood, etc.
* 5 Subjects of childbearing age agree to take effective contraceptive measures throughout the trial period, and continue to 28 days after the last medication.
* 6 Volunteer to participate in this study, sign an informed consent form, have good compliance, and be able to cooperate with the experimental observation.

Exclusion Criteria:

* 1 Any other bleeding disease except Congenital hemophilia A or B.
* 2 Patients with any previous medical history or symptoms of arterial or venous thromboembolic events (such as atherosclerosis, myocardial infarction, ischemic stroke, transient ischemic attack, deep vein thrombosis or pulmonary hypertension embolism) or disseminated intravascular coagulation (DIC) within the past 1 year.
* 3 Baseline and previous values of FⅦ inhibitor or activated recombinant human coagulation factor VII inhibitor is positive.
* 4 Vitamin K deficiency.
* 5 Human immunodeficiency virus (HIV) positive and cluster of differentiation 4 (CD4) count ≤200/μl, the number of virus carriers ≥200 particles/μl or ≥400000 copies/ml.
* 6 Subjects plan to perform elective surgery during the trial period.
* 7 Those who are allergic to test drugs or any excipients.
* 8 Severe anemia and need blood transfusion.
* 9 Platelet count <80×10^9/L.
* 10 Obvious liver or kidney damage: glutamic-pyruvic transaminase (ALT) or aspartic transaminase (AST)>2.5×ULN, or total bilirubin>1.5×ULN or serum creatinine>1.5×ULN.
* 11 Severe heart disease, including myocardial infarction, cardiac insufficiency grade 3 or above, the current New York Heart Association cardiac function grade II-IV.
* 12 There was a prior intracranial hemorrhage
* 13 Those who had used or planned to use any anticoagulants, antifibrinants and drugs affecting platelet function during the first week of medication included non-steroidal anti-inflammatory drugs (NSAIDs) such as aspirin
* 14 Hypertension that cannot be controlled with drug treatment: systolic blood pressure> 150 mmHg or diastolic blood pressure> 90 mmHg.
* 15 Participated in other clinical studies (except Activated coagulation factor VII, coagulation factor VIII and coagulation factor IX trials) within one month before the first medication.
* 16 Alcoholism, drug abuse, mental disorders, other severe acute or chronic diseases, greater abnormal laboratory values, and those who are considered unsuitable by the researcher.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Number of bleeding Effective rate of hemostasis | Each new blood event was assessed within 12 hours of initial treatment
  Hemostasis is effective after the bleeding event if the bleeding event has not received other treatment within 12 hours since the first treatment and achieved moderate or above remission (based on the four-point scoring standard)
Activity recovery of first dose | Within 1 hour of completion of infusion
  The peak coagulation factor VII activity measured within 1 hour after the end of the infusion was subtracted from the baseline coagulation factor VII activity and expressed as [IU/ml]/[IU/kg].

SECONDARY OUTCOMES:
Number of bleeding effective rate of hemostasis within 8 hours | Each new blood event was assessed within 8 hours of initial treatment
  Excellent remission (based on the four-point scoring standard)
Number of bleeding effective rate continuous hemostatic | Each new blood event was assessed within 24 hours of initial treatment
  Moderate or above remission (based on grade 4 scoring criteria) without receiving other treatment within 24 hours after the occurrence of bleeding event is considered as effective hemostasis after the occurrence of bleeding event.
Activity recovery after repeated administration | Within 1 hour of completion of infusion
  The peak coagulation factor VII activity measured within 1 hour after the end of the infusion was subtracted from the baseline coagulation factor VII activity and expressed as [IU/ml]/[IU/kg].
Dose of injections for each new blood transfusion | Up to 24 weeks.
  Dose of injections for each new blood transfusion.The dose of injections (including average injection dose and total dose) of each new blood transfusion were recorded.
Number of injections for each new blood transfusion | Up to 24 weeks.
  Number of injections for each new blood transfusion.The number of injections of each new blood transfusion were recorded.
Coagulation tests | First and week 24, within 30 minutes before the administration and 5 minutes after the completion of drug injection.
  Coagulation tests: Changes of activated partial thromboplastin time (APTT).
Coagulation tests | First and week 24, within 30 minutes before the administration and 5 minutes after the completion of drug injection.
  Coagulation indicators: Changes of prothrombin time (PT).
Coagulation tests | First and week 24, within 30 minutes before the administration and 5 minutes after the completion of drug injection.
  Coagulation indicators: Changes of thrombin time(TT).
Coagulation tests | First and week 24, within 30 minutes before the administration and 5 minutes after the completion of drug injection.
  Coagulation indicators: Changes of fibrinogen (Fbg).
Coagulation tests | First and week 24，within 30 minutes before the administration and 5 minutes after the completion of drug injection.
  Coagulation indicators: thrombin production test (TGA):Changes of thrombin production potential (ETP) in TGA at each test time.

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Affiliated Hospital of North China University of Science and Technology, Tangshan, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Hematology Hospital of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality